CLINICAL TRIAL: NCT05880186
Title: Influence of the Time of Day in the Effect of Caffeine on Maximal Fat Oxidation During Exercise in Women. A Randomized, Crossover, Double-blind, and Placebo-controlled Study
Brief Title: Influence of the Time of Day in the Effect of Caffeine on Maximal Fat Oxidation During Exercise in Women
Acronym: CIRCAF_WOM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Francisco de Vitoria (Other)
Collaborators: Universidad de Granada (Other); Universidad Rey Juan Carlos (Other); Camilo Jose Cela University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UFVitoria_2
Record Dates: First submitted 2023-05-18; First posted 2023-05-30 (Actual); Last update posted 2023-05-30 (Actual); Status verified 2023-05

CONDITIONS: Dietary Supplement

STUDY DESIGN:
Intervention Model Description: Dietary Supplement: caffeine acute supplementation
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Caffeine intake (Experimental): Test in the morning
  A dose of 3 mg/kg of caffeine (Bulk Powders, Essex, United Kingdom) was ingested before the beginning of each test.
  Test in the evening
  A dose of 3 mg/kg of caffeine (Bulk Powders, Essex, United Kingdom) was ingested before the beginning of each test.
  Interventions: Dietary Supplement: Acute caffeine supplementation
- Placebo intake (Placebo Comparator): Test in the morning
  A dose of 3 mg/kg of placebo (Cellulose, Guinama, Valencia, Spain) was ingested before the beginning of each test.
  Test in the evening
  A dose of 3 mg/kg of placebo (Cellulose, Guinama, Valencia, Spain) was ingested before the beginning of each test
  Interventions: Dietary Supplement: Acute caffeine supplementation

INTERVENTIONS:
Dietary Supplement: Acute caffeine supplementation — To evaluate the influence of the time of the day (i.e., morning vs evening) on the effect of caffeine on maximal fat oxidation in women.

SUMMARY:
Caffeine is a natural stimulant with well-recognized metabolic benefits, however, there is a lack of studies investigating the time-of-day caffeine influence to enhance fat oxidation in women. The aim of this study was to evaluate the influence of the time of the day on the effect of caffeine on maximal rate of fat oxidation during aerobic exercise in women.

DETAILED DESCRIPTION:
Caffeine is a natural stimulant with well-recognized sports performance benefits. Aside its performance-enhancing effect, caffeine has the potential of increasing fat utilization during aerobic exercise at submaximal intensities, lowering-down the contribution of carbohydrate as a fuel. This property of caffeine may provoke a glycogen-sparing effect in the skeletal muscle and liver for exercise situations where carbohydrate availability may be a challenge. Additionally, the capacity of caffeine to enhance fat utilization during exercise could be of interest for improving health outcomes as it may increase the rate of change in body composition in exercise programs. Maximal fat oxidation rate (MFO) during exercise is a remarkable physiological indicator associated with metabolic flexibility/body weight loss and endurance performance To date, it is unknown if caffeine increases MFO in the same proportion during morning and evening exercise trials in women. For this reason, the aim of the present study was to evaluate the influence of the time of the day on the effect of caffeine on MFO in women. We hypothesised that caffeine would increase MFO during morning and evening exercise and this effect would be of similar magnitude at both times of day.

ELIGIBILITY:
Inclusion Criteria:

* To be non-smokers.
* To have low caffeine intake (i.e., < 50 mg of caffeine per day in the previous 2 months)
* To show no previous history of cardiopulmonary diseases or having suffered musculoskeletal injuries in the previous 6 months.
* To have a regular duration of their menstrual cycle for the previous 6 months.
* To confirm no existence of any type of menstrual disorders such as dysmenorrhea, amenorrhea, or strong symptoms associated with pre-menstrual syndrome.

Exclusion Criteria:

-

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2021-02-09 (Actual); Primary Completion 2021-04-09 (Actual); Study Completion 2021-04-09 (Actual)

PRIMARY OUTCOMES:
MFO | 2-months
  Maximal fat oxidation during exercise

SECONDARY OUTCOMES:
FATmax | 2-months
  The intensity of exercise that elicits MFO
RPE | 2-months
  Rate of percevied exertion during exercise
FAT AND CHO oxidation | 2-months
  Fat and carbohydrates oxidation

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Francisco de Vitoria, Pozuelo de Alarcón, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Munoz A, Aguilar-Navarro M, Ruiz-Moreno C, Varillas-Delgado D, Amaro-Gahete FJ, Gutierrez-Hellin J, Del Coso J, Lopez-Samanes A. Influence of the time of day in the effect of caffeine on maximal fat oxidation during exercise in women: a randomized, crossover, double-blind, and placebo-controlled study. Eur J Appl Physiol. 2024 Mar;124(3):849-859. doi: 10.1007/s00421-023-05312-2. Epub 2023 Sep 20. PMID 37728787